CLINICAL TRIAL: NCT03528902
Title: Tamoxifen Therapy to Treat Pulmonary Arterial Hypertension
Acronym: T3PAH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Eric Austin, Associate Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 180241
Record Dates: First submitted 2018-03-21; First posted 2018-05-18 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Hypertension; Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension; Primary Pulmonary Hypertension; Lung Diseases; Tamoxifen; Estrogen Receptor Antagonist; Hormone Antagonists; Estrogens
MeSH Terms: conditions — Hypertension; Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension; Lung Diseases | interventions — Tamoxifen

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, double-blind, placebo-controlled Phase II study of 24 subjects with PAH. Eligible subjects will be randomized to treatment with a 1:1 ratio using a permuted-block randomization algorithm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamoxifen (Experimental): 20 mg po TID for 24 weeks
  Interventions: Drug: Tamoxifen
- Placebo (Placebo Comparator): Placebo arm
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Tamoxifen — Tamoxifen 20 mg po daily for 24 weeks.
  Arms: Tamoxifen
Drug: Placebo Oral Tablet — Placebo
  Arms: Placebo

SUMMARY:
The main purpose of this clinical trial is to examine the feasibility and effects of tamoxifen in subjects with pulmonary arterial hypertension (PAH). The study will evaluate how well the drug is tolerated, and its impact on functional condition and selected biomarkers. Changes in tricuspid annular plane systolic excursion (TAPSE) and other parameters determined by transthoracic echocardiography will be evaluated as well as changes in additional metrics such as six minute walk test distance, quality of life assessments, and hormone levels.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is characterized by progressive loss of function by the pulmonary vascular bed due to a variety of factors including obliterative vascular lesions, vasoconstriction, and thrombotic occlusion of the pulmonary arteries. Ultimately, right-sided heart failure ensues with severe limitation of exercise and eventual progression to death or lung transplantation. While there are multiple FDA-approved therapies for PAH representing 3 major pathways of interest, no treatments are curative, and have additional limitations including high expense, multiple side effects, and dosing inconveniences.

The strongest established risk factor for the progressively fatal disease pulmonary arterial hypertension (PAH) is female sex (~3:1 female:male ratio). We and others have found higher circulating estrogen levels, and enhanced estrogen signaling, in PAH patients. Preclinical work by our group and others supports the concept that anti-estrogen therapy, is effective for both prevention and treatment in PAH. Recent and ongoing clinical studies are underway to assess these approaches in humans, including a recent study demonstrating the safety of estrogen reduction in postmenopausal women.

Tamoxifen is the most commonly used selective estrogen receptor modulator (SERM). Due to its extensive use in humans for over three decades, it has an excellent safety profile and its long-term sequelae are well characterized. Furthermore, it is a generic drug which has been FDA-approved for treatment and prevention of breast cancer, particularly those with estrogen receptor-positive neoplasms.

To help to determine whether tamoxifen may be a safe and effective treatment for PAH in women and men, we will conduct a single-center, randomized, double-blind, placebo-controlled Phase II study of subjects with PAH. All subjects will also be treated with background standard of care therapy at the discretion of their PAH care physician.

ELIGIBILITY:
Inclusion Criteria:

* Previous documentation of mean pulmonary artery pressure greater than or equal to 25 mm Hg with a pulmonary capillary wedge pressure (or left ventricular end-diastolic pressure) less than or equal to15 mm Hg and PVR greater than or equal to 3 WU at any time before study entry, consistent Group 1 PAH classified by accepted international classification.
* Diagnosis of PAH which is idiopathic, heritable, drug- or toxin-induced, or associated with connective tissue disease.
* Age 18 years and older.
* WHO Functional Class I, II, or III status.
* Ability to perform a six minute walk test without significant limitations in musculoskeletal function or coordination, with distance greater than or equal to 150m and less than or equal to 550m.
* Informed consent.

Exclusion Criteria:

* Current treatment with estrogen, progesterone, or any form of sex hormone therapy.
* Current treatment with anti-sex hormone therapy (e.g., anastrozole, fulvestrant, tamoxifen, leuprolide acetate (luporon) or other centrally-acting hormone agents.
* WHO Functional Class IV status.
* History of, or current, breast, uterine, ovarian, or testicular cancer.
* Current pregnancy, or prior pregnancy within 3 months of enrollment.
* Initiation of PAH therapy (prostacyclin analogues, endothelin-1 receptor antagonists, phosphodiesterase-5 inhibitors, riociguat, selexipag) within three months of enrollment; the dose must be stable for at least three months prior to Baseline Visit. Of note, PAH therapy, including diuretics, which is stopped and then restarted or has dose changes which are not related to initiation and up titration will be allowed within 3 months prior to the Baseline Visit, and during the trial for subjects.
* History of thromboembolic event.
* Hospitalized or acutely ill.
* Renal failure (creatinine over 2.0).
* Hypercalcemia.
* Severe osteoporosis (t score < -2.0 OR t score < -2.5 if on bone modifying treatment).
* Current or recent (< 3 months) chronic heavy alcohol consumption.
* Enrollment in a clinical trial or concurrent use of another investigational drug (non FDA approved) or device therapy within 30 days of screening visit.
* Enrollment in any pharmacologic clinical trial within one month of screening.
* Due to potential drug interactions with tamoxifen, subjects using bosentan (CYP3A4) or selexipag (CYP2C8) will be excluded.
* Due to the concerns of pregnancy during PAH and with tamoxifen use, subjects will be excluded who do not use at least two forms of contraception (e.g., IUD plus the use of a barrier contraceptive method).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Since the data that will be produced involves patients with a disease process that is much in need of new treatment options and the investigators agree that data sharing is essential for expedited translation of research results into patient treatment options. A detailed data sharing plan is in place and available upon request. In brief:
  It is our plan to make data available at the time it is accepted for publication of the main findings from the final dataset through the use of a data enclave of our own design that would restrict our Data Analyst from sharing any information that would breach participant confidentiality. Potential researchers will contact the PI to discuss specific needs and how the data will be utilized. A formal approval process is in place to evaluate and complete such requests.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 2 years after study completion.
Access Criteria: Criteria include:
  * detailed written description of the project for which the data would be used.
  * acknowledge in any publication resulting from the data, the source of the data, crediting the program support.
  * agree to submit all papers or reports submitted for publication to the PI for review prior to submission.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between 1/08/2018-12/28/2022
Groups:
- Placebo: Placebo arm
  Placebo Oral Tablet: Placebo daily for 24 weeks.
Period: Overall Study
Arm/Group | Tamoxifen | Placebo
Started | 9 | 9
Completed | 8 | 9
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamoxifen | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (12.4) | 51 (10.5) | 48.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Transthoracic Echocardiogram (ECHO)-Based Change in the Tricuspid Annular Plane Systolic Excursion (TAPSE) Measurement
Description: Transthoracic echocardiograms (ECHOs) will be performed to measure the TAPSE value prior to Intervention at Week 0, as well as at the end of the study intervention (Week 24). The primary outcome measure will be the change in TAPSE, determined by echocardiogram, from Week 0 to Week 24.
  About TAPSE: Tricuspid annular plane systolic excursion (TAPSE) is a parameter of global right ventricular function which describes apex-to-base shortening of the ventricle. It is obtained by transthoracic echocardiogram, which can be performed on a resting subject without sedation in the outpatient setting. TAPSE correlates closely with the right ventricular ejection fraction, and has been determined to be both highly specific and easy to measure.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 8 | 8
mm
  Baseline | 2.244 (0.194) | 2.244 (0.274)
  Week 24 | 2.300 (0.220) | 2.212 (0.352)

2. Secondary Outcome: Six Minute Walk Test Distance (6MWTD)
Description: Change in 6MWTD from Week 0 to Week 24. The 6-minute walk test distance (6MWTD) is a widely accepted measure of exercise capacity and functional status. The 6MWTD is a clinical and research test obtained in a standardized manner according to American Thoracic Society (ATS) Guidelines.
  Briefly, the 6MWT is a sub-maximal exercise test on flat ground that is used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity over time.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 8 | 8
Meters
  Baseline | 375.3 (78.4) | 415.2 (87.5)
  Week 24 | 377.9 (84.5) | 405.5 (156.4)

3. Secondary Outcome: Quality of Life Will be Assessed Using the SF36 Questionnaire. This Will be Administered at Baseline and 12 and 24 Weeks.
Description: Change in score from Week 0 to Week 24.
  Specifically, Quality of life will be assessed using two different accepted questionnaires for pulmonary hypertension patients, the SF36 questionnaires. These will be administered at baseline and 12 and 24 weeks. Note that all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 9 | 9
score on a scale
  physical_functioning (Baseline) | 55 [35 to 55] | 65 [45 to 85]
  physical_health(Baseline) | 31.2 [12.5 to 62.5] | 81.2 [50 to 93.8]
  emotional_probs (Baseline) | 66.67 [25 to 91.67] | 100 [91.67 to 100]
  energy_fatigue (Baseline) | 37.5 [18.8 to 62.5] | 62.5 [50 to 75]
  well_being (Baseline) | 75 [60 to 90] | 90 [85 to 100]
  social_function (Baseline) | 62.5 [50 to 87.5] | 100 [87.5 to 100]
  pain (Baseline) | 67.5 [45 to 90] | 67.5 [60 to 90]
  gen_health(Baseline) | 40 [35 to 45] | 50 [35 to 65]
  physical_functioning (Week 24) | 55 [38.8 to 72.5] | 65 [55 to 78.6]
  physical_health (week 24) | 40.6 [28.1 to 50] | 93.8 [50 to 100]
  emotional_probs (Week 24) | 58.3 [50 to 100] | 100 [100 to 100]
  energy_fatigue (Week 24) | 59.4 [45.3 to 81.2] | 62.5 [50 to 81.2]
  well_being (Week 24) | 77.5 [68.8 to 92.5] | 90 [65 to 90]
  social_function (Week 24) | 81.2 [50 to 100] | 100 [62.5 to 100]
  pain (Week 24) | 67.5 [51.9 to 77.5] | 77.5 [45 to 90]
  gen_health (Week 24) | 37.5 [28.8 to 56.2] | 40 [35 to 70]

4. Secondary Outcome: Quality of Life Will be Assessed Using emPHasis-10 Questionnaire. This Will be Administered at Baseline and 12 and 24 Weeks.
Description: This will be administered at baseline and 12 and 24 weeks. Change in score from Week 0 to Week 24 will be reported. emPHasis-10 scores range from 0 to 50, higher scores indicate worse quality of life
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 8 | 9
units on a scale
  Baseline | 25.7 (13.9) | 14.3 (11.7)
  Week 24 | 23.5 (12.7) | 15.9 (13.7)

5. Other Pre Specified Outcome: Plasma BNP
Description: Change in Plasma BNP levels will be assessed from Week 0 to Week 24 during the study. These measurements are made from the plasma, and will require a blood draw from the research participant.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 8 | 8
pg/mL
  Baseline | 30.4 (31.3) | 79.1 (110.5)
  Week 24 | 101.3 (150.9) | 76.2 (77.1)

6. Other Pre Specified Outcome: HgbA1c
Description: Change in hemoglobin A1c (HgbA1c) levels will be assessed from Week 0 to Week 24 during the study. These measurements are made from the plasma, and will require a blood draw from the research participant.
Time Frame: 24 weeks
Population: HgbA1c was not assessed due to assay issues.
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were monitored throughout the duration of enrollment but were specifically reviewed with participants at weeks 3, 6, 9, 12, 15, 18, 21 and 24.
Arm/Group | Tamoxifen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 2/9
Other Adverse Events (participants affected / at risk) | 5/9 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamoxifen (N=9) | Placebo (N=9)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamoxifen (N=9) | Placebo (N=9)
Hot Flashes (General disorders) | 3 (3) | 1 (1)
Night Sweats (General disorders) | 1 (1) | 2 (4)
Mood Alterations (Psychiatric disorders) | 1 (1) | 2 (2)
Nonspecific pain (General disorders) | 1 (1) | 0 (0)
Alteration in smell (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT03528902/Prot_SAP_000.pdf